CLINICAL TRIAL: NCT02521051
Title: A Phase I/II Trial to Evaluate the Safety and Tolerability of Alectinib and Bevacizumab in Patients With Advanced, ALK-Positive, Non-Small Cell Lung Cancer
Brief Title: Phase I/II Trial of Alectinib and Bevacizumab in Patients With Advanced, Anaplastic Lymphoma Kinase (ALK)-Positive, Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Justin Gainor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-055
Record Dates: First submitted 2015-07-20; First posted 2015-08-13 (Estimated); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer (NSCLC); Anaplastic lymphoma kinase; ALK; Brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — alectinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg (Experimental): Participants were administered Alectinib 600 mg twice daily by mouth, and Bevacizumab 15 mg/kg intravenously once every 3 weeks. DLTs will be monitored and evaluated throughout the first cycle (21 days).
  Interventions: Drug: Alectinib; Drug: Bevacizumab
- Phase I Dose Level -1: Alectinib 600 mg + Bevacizumab 7.5 mg/kg (Experimental): Participants were administered Alectinib 600 mg twice daily by mouth, and Bevacizumab 7.5 mg/kg intravenously once every 3 weeks. DLTs will be monitored and evaluated throughout the first cycle (21 days).
  Interventions: Drug: Alectinib; Drug: Bevacizumab
- Phase I Dose Level -2: Alectinib 450 mg + Bevacizumab 7.5 mg/kg (Experimental): Participants were administered Alectinib 450 mg twice daily by mouth, and Bevacizumab 7.5 mg/kg intravenously once every 3 weeks. DLTs will be monitored and evaluated throughout the first cycle (21 days).
  Interventions: Drug: Alectinib; Drug: Bevacizumab
- Phase II: RP2D (Experimental): In the phase II portion of the study, all patients received alectinib plus bevacizumab at the RP2D determined in the phase I portion.
  Interventions: Drug: Alectinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Alectinib
  Other Names: Alecensa
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
This research study is evaluating two drugs, alectinib and bevacizumab, as possible treatments for Advanced Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial.

* A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose(s) of the investigational intervention to use for further studies.
* Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease.
* "Investigational" means that the intervention is being studied.

  * In this research study, the investigators are investigating the combination of two study drugs: alectinib and bevacizumab. The FDA (the U.S. Food and Drug Administration) has not approved alectinib as a treatment for any disease.

It has been found that some people with NSCLC have a change (mutation) in a certain gene called the anaplastic lymphoma receptor tyrosine kinase (ALK) gene. This mutated gene helps cancer cells grow.

-- Alectinib belongs to a class of drugs designed to inhibit ALK. This drug has been used in other research studies. Information from those other research studies suggests that alectinib may be effective in killing cancer cells that have changes in ALK. Only participants with changes in the ALK gene will be allowed to participate in this study.

In this research study, Alectinib will be combined with Bevacizumab. -- Bevacizumab (also called Avastin) works by slowing or stopping the growth of cells in cancer tumors by decreasing the blood supply of the tumors. If blood supply is decreased, oxygen and nutrients that are needed for tumor growth are decreased. The FDA has approved Bevacizumab as a treatment option for your disease

The purpose of this study is to test the safety of Alectinib and Bevacizumab. The investigators will also determine how effective this combination is in participants with advanced, ALK-positive NSCLC with a focus on participants with brain metastases.

In the phase I portion of the study, a 3 + 3 dose de-escalation design was to determine the recommended phase II dose (RP2D) of alectinib and bevacizumab. Three patients will be treated per cohort for one cycle (21 days per cycle) beginning with dose level 1 cohort.

* Dose level 1 (starting dose) = Alectinib 600mg twice daily orally (PO), and Bevacizumab 15 mg/kg administered intravenously (IV) every 3 weeks.

  -- Dose level 1 was selected based on the individual RP2Ds for each medication and anticipation for minimal overlapping toxicities.
* Dose level -1 = Alectinib 600mg twice daily orally (PO),and Bevacizumab 7.5 mg/kg administered intravenously (IV) every 3 weeks.
* Dose level -2 = Alectinib 450mg twice daily orally (PO), and Bevacizumab 7.5 mg/kg administered intravenously (IV) every 3 weeks.

DLTs were defined as adverse events (AEs) occurring within the first cycle of treatment (21 days) attributed to the study drugs, and grade 3 or higher according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. If no DLTs are observed with dose level 1 cohort, we will enroll an additional 3 participants (6 total) to the same cohort and proceed with the phase II portion of the study if one or less experience a DLT. In any other dose level cohort, if one of three patients experiences a DLT, another 3 patients will be treated at the same dose level for one cycle. If no additional DLTs are observed, we will proceed with the phase II portion of the trial. If more than one of 3 patients develops a DLT in any cohort, another 3 patients will be treated in the next lowest dose cohort.

The RP2D for the combination of alectinib and bevacizumab was defined as either (i) the highest dosage cohort in which less than a third of patients experienced a DLT, or (ii) alectinib at the previously defined RP2D as a single agent (600 mg twice daily) plus bevacizumab at the highest tolerated dose investigated for the indication (15 mg/kg every 21 days), whichever was the lower dose.

In the phase II portion of the study, all patients received alectinib plus bevacizumab at the RP2D determined in the phase I portion. Cycles were 21 days long. Treatment was continued until there was evidence of progressive disease, death, or unacceptable toxicity. Patients were allowed to continue study drugs beyond progression if deemed clinically beneficial at the investigator's discretion. Intra-patient dose modification of bevacizumab was not permitted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced, non-squamous, non-small cell lung cancer.
* Molecular confirmation of an ALK rearrangement.
* Age ≥ 18 years old.
* Life expectancy > 12 weeks.
* Performance status 0-2.
* Adequate hematologic function:
* Adequate renal function:

  * An estimated Glomerular Filtration Rate (eGFR) of at least 45 mL/min/1.73 m2
  * International normalized ration (INR)≤ 1.5
  * Partial thromboplastin time (PTT) ≤1.5 x upper limit of normal (ULN)
* For all females of childbearing potential, a negative pregnancy test must be obtained within 3 days before starting study treatment.
* Able and willing to provide written informed consent
* Phase II Only:
* Presence of at least one measurable central nervous system (CNS) target lesion (At least 5 mm in size)

  * Lesions must be untreated or progressive according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after previous local therapy.
  * Participants who are receiving corticosteroids must be on a stable or decreasing dose
* At least one measurable extra-CNS lesion based upon RECIST version 1.1.

Exclusion Criteria:

* Squamous cell histology or mixed, predominantly squamous adenosquamous carcinoma
* Previous history of haemoptysis
* Tumour infiltrating into large vessels or infiltrating into the proximal tracheobronchial network
* Unstable, symptomatic brain metastases.
* History of hemorrhagic CNS metastases
* History of intracranial hemorrhage (either by clinical history or neuroimaging)
* History of or genetic predisposition to a bleeding diathesis or coagulopathy
* Therapeutic anticoagulation
* Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325 mg/day)
* Clinically significant heart disease (i.e., active), stroke or myocardial infarction within 6 months prior to enrolment, unstable angina pectoris, congestive heart failure of grade > II according to the New York Heart Association (NYHA), or cardiac arrhythmia requiring specific treatment
* Arterial or venous thromboembolic events within 6 months of study enrollment.
* Poorly controlled arterial hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg)
* Invasive surgical intervention within 28 days prior to the start of treatment
* Minor surgical intervention, including placement of a permanent catheter within 24 hours prior to the first infusion of bevacizumab.
* Non-healing wound, active peptic ulcer or bone fracture.
* Previous history of abdominal fistula, tracheoesophageal fistula or other fistula with grade 4 severity, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to enrolment.
* Proteinuria at baseline.
* Previous anti-angiogenic treatment
* Patients previously treated with alectinib (Phase II only).
* Radical radiotherapy to the thorax with curative intent within 28 days
* Cytotoxic chemotherapy within 21 days prior to enrolment.
* Treatment with crizotinib within 7 days prior to enrolment. For all other ALK Tyrosine kinase inhibitors (TKIs), the washout period should be ≥5 half-lives prior to enrolment.
* Any GI disorder that may affect absorption of oral medications
* Alanine transaminase (ALT) or aspartate transaminase (AST) > 3 × ULN (≥5 × ULN for patients with concurrent liver metastasis)
* Impaired excretory function (e.g., hyperbilirubinemia) or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices
* Acute viral or active autoimmune, alcoholic, or other types of hepatitis
* National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (version 4.0) Grade 3 or higher toxicities due to any prior therapy (e.g. radiotherapy) (excluding alopecia),
* History of organ transplant.
* Co-administration of anti-cancer therapies other than those administered in this study.
* QTc > 470 ms or patients with symptomatic bradycardia.
* Administration of strong/potent cytochrome P450 (CYP)3A inhibitors or inducers within 14 days
* Administration of agents with potential QT interval prolonging effects within 14 days prior to the first administration of study drug and while on treatment.
* History of hypersensitivity to any of the additives in the alectinib drug formulation
* Documented allergy or hypersensitivity to monoclonal antibodies (bevacizumab)
* History of drug-induced pneumonitis or hypersensitivity pneumonitis from prior ALK TKI therapy.
* Pregnant or lactating women.
* Known HIV positivity or AIDS-related illness.
* Any condition or illness that could compromise patient safety or interfere with the evaluation of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gainor, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase I Dose Level -1: Alectinib 600 mg + Bevacizumab 7.5 mg/kg | Phase I Dose Level -2: Alectinib 450 mg + Bevacizumab 7.5 mg/kg | Phase II: RP2D
Started | 6 | 0 | 0 | 5
Completed | 6 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 42 [32 to 64] | 50 [25 to 66] | 46 [25 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  Never | 5 | 3 | 8
  Light (less than 10 pack-years) | 1 | 2 | 3
Brain metastases [Count of Participants; unit: Participants]
  Present | 4 | 5 | 9
  Absent | 2 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG performance score assesses a participant's level of function and capability of self-care. Scores range from 0 to 5, with higher scores indicating lower levels of function. Study eligibility criteria allowed participants with ECOG scores 0-2 to be enrolled.
  * Score 0 = Fully active, asymptomatic.
  * Score 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  * Score 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, in bed <50% of waking hours
  Participants
    Score 0 | 4 | 3 | 7
    Score 1 | 1 | 2 | 3
    Score 2 | 1 | 0 | 1
Prior anaplastic lymphoma kinase (ALK) tyrosine kinase inhibitor (TKI) therapy [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: (Phase 1) Recommended Phase II Dose of Alectinib
Description: The recommended phase II doses for the combination of alectinib and bevacizumab will be defined as either a) the highest dosage cohort in which less than 1/3 of patients experience a dose-limiting toxicity or b) alectinib at the previously defined recommended phase II dose (600 mg twice daily PO) as a single agent plus bevacizumab at the highest tolerated dose (15 mg/kg IV every 21 days) investigated in this indication - whichever is the lower dose.
  Dose-limiting toxicities (DLTs) were defined as adverse events (AEs) occurring within the first cycle of treatment (21 days) attributed to the study drugs.
Time Frame: first cycle of treatment (21 days)
Measure: Number; unit: mg
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg
Number analyzed (Participants) | 6
mg | 600

2. Primary Outcome: (Phase 1) Recommended Phase II Dose of Bevacizumab
Description: as for outcome 1
Time Frame: first cycle of treatment (21 days)
Measure: Number; unit: mg/kg
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg
Number analyzed (Participants) | 6
mg/kg | 15

3. Primary Outcome: (Phase 2) Number of Participants With Intracranial Hemorrhagic Events Who Received RP2D
Description: In the phase II portion of the study, we aim to further investigate the safety and tolerability of alectinib plus bevacizumab at the RP2Ds as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The combination of alectinib and bevacizumab will be deemed unsafe if 2 or more participants are observed to have grade 2 or higher, central nervous system (CNS) intracranial hemorrhagic events.
Time Frame: up to 4 years
Population: RP2Ds for alectinib plus bevacizumab were confirmed in August 2016. Enrollment for the phase II cohort occurred from August 2016 to February 2020. We initially planned to enroll 20 participants to the phase II cohort but due to slow accrual, the decision was made to stop the study prematurely in July 2021.
Measure: Number; unit: participants
Arm/Group | Phase II: RP2D
Number analyzed (Participants) | 5
participants | 0

4. Secondary Outcome: Central Nervous System Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with complete response (CR) or partial response (PR), evaluated using a modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria for CNS response:
  * CR = Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to less than 10 mm.
  * PR = At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 6 | 5
percentage of participants | 66.66 | 60.00

5. Secondary Outcome: Central Nervous System Disease Control Rate
Description: Disease control rate (DCR) is the percentage of participants with intracranial complete response (CR), partial response (PR), and stable disease (SD), evaluated using a modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria for CNS response:
  * CR = Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to less than 10 mm.
  * PR = At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters.
  * SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the baseline sum diameters.
  * PD = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters. At least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions also qualifies as PD.
Time Frame: Up to 4 years
Population: One participant from the phase 1 cohort was excluded from analysis because they didn't have an intracranial lesion(s) at enrollment, nor did they develop any while on study.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 5 | 5
percentage of participants | 100 | 100

6. Secondary Outcome: Central Nervous System Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from the start of study treatment to the date of progressive disease (PD) in the central nervous system (CNS) or death due to CNS disease. PD is evaluated using a modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria for CNS response:
  * PD = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters. At least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions also qualifies as PD.
Time Frame: up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 6 | 5
months | 23.87 [10.36 to 40.52] | 7.21 [3.44 to 27.51]

7. Secondary Outcome: Overall Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with intra- and extra-cranial complete response (CR) or partial response (PR), evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1.
  * CR = Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to less than 10 mm.
  * PR = At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 6 | 5
percentage of participants | 83.33 | 60.00

8. Secondary Outcome: Overall Disease Control Rate
Description: Disease control rate (DCR) is the percentage of participants with intra- and extra-cranial complete response (CR), partial response (PR), and stable disease (SD), evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version1.1:
  * CR = Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to less than 10 mm.
  * PR = At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters.
  * SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the baseline sum diameters.
  * PD = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters. At least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions also qualifies as PD.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 6 | 5
percentage of participants | 100 | 100

9. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from the start of study treatment to the date of progressive disease (PD) or death due to any cause. PD is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version1.1:
  - PD = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum diameters. At least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions also qualifies as PD.
Time Frame: up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 6 | 5
months | 23.64 [9.02 to 40.52] | 4.95 [4.26 to 27.51]

10. Secondary Outcome: Health-related Quality of Life Questionnaire EORTC QLQ-C30
Description: The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of functional scales, symptom scales, a global health status/quality of life (QOL) scale. All of the scales range in score from 0 to 100. A summary score is calculated as the average of all scores. High score for functional scales mean high level of functioning. High score for global health status means high quality of life. High score for symptom scales mean high level of problems.
Time Frame: Baseline to cycle 7 (21 weeks)
Population: Only participants who completed the baseline questionnaire and C7D1 post-treatment questionnaire will be included in the analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 2 | 1
score on a scale
  Baseline: Functional scales | 86.67 [77.78 to 95.56] | 42.22 [NA to NA] — not applicable for a single participant
  Cycle7: Functional scales | 87.78 [82.22 to 93.33] | 68.89 [NA to NA] — not applicable for a single participant
  Baseline: Symptom scales | 15.38 [12.83 to 17.95] | 38.46 [NA to NA] — not applicable for a single participant
  Cycle7: Symptom scales | 12.83 [7.69 to 17.94] | 30.77 [NA to NA] — not applicable for a single participant
  Baseline: Global health status/QOL | 75.00 [66.67 to 83.33] | 25.00 [NA to NA] — not applicable for a single participant
  Cycle7: Global health status/QOL | 58.33 [50 to 66.67] | 75.00 [NA to NA] — not applicable for a single participant

11. Secondary Outcome: Health-related Quality of Life Questionnaire Specific to Brain Cancer: EORTC QLQ-BN20
Description: The European Organization for Research and Treatment of Cancer quality of life questionnaire has a brain cancer nodule (EORTC QLQ-BN20) developed for patients undergoing chemotherapy or radiotherapy. It includes 20 items, 13 of which aggregate into four scales assessing future uncertainty, visual disorder, motor dysfunction, and communication deficit. The remaining single items assess other disease symptoms (e.g. headaches and seizures) and treatment toxic effects (e.g. hair loss). Raw scores items were computed and subsequently transformed linearly to a 0-100 scale. A higher score represents worse quality of life.
Time Frame: Baseline, Cycle 7 Day 1 (21 weeks)
Population: Only participants who completed the baseline questionnaire and C7D1 questionnaire will be included in the analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
Number analyzed (Participants) | 3 | 1
score on a scale
  Baseline: Future uncertainty | 38.89 [0.00 to 66.67] | 58.33 [NA to NA] — not applicable for a single participant
  Cycle7: Future uncertainty | 16.67 [0 to 33.33] | 33.33 [NA to NA] — not applicable for a single participant
  Baseline: Visual disorder | 7.41 [0.00 to 22.22] | 0.00 [NA to NA] — not applicable for a single participant
  Cycle7: Visual disorder | 0.00 [0.00 to 0.00] | 0.00 [NA to NA] — not applicable for a single participant
  Baseline: Motor dysfunction | 0.00 [0.00 to 0.00] | 22.22 [NA to NA] — not applicable for a single participant
  Cycle7: Motor dysfunction | 0.00 [0.00 to 0.00] | 11.11 [NA to NA] — not applicable for a single participant
  Baseline: Communication deficit | 0.00 [0 to 0] | 77.78 [NA to NA] — not applicable for a single participant
  Cycle7: Communication deficit | 0.00 [0.00 to 00.00] | 100.00 [NA to NA] — not applicable for a single participant
  Baseline: other symptoms | 9.52 [0 to 19.05] | 19.05 [NA to NA] — not applicable for a single participant
  Cycle7: other symptoms | 15.87 [9.52 to 28.57] | 19.05 [NA to NA] — not applicable for a single participant

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg | Phase II: RP2D
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg (N=6) | Phase II: RP2D (N=5)
Hypertension (Vascular disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: Alectinib 600 mg + Bevacizumab 15 mg/kg (N=6) | Phase II: RP2D (N=5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Fatigue (General disorders) | 5 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 1
Hypertension (Vascular disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2
Edema limbs (General disorders) | 2 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
CPK increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Bilirubin increased (Investigations) | 2 | 2
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Hemoptysis
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 — gingival bleeding
Hematoma (Vascular disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 — tongue sensitivity
Headache (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — sinus congestion
Palpitations (Cardiac disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Flu-like symptoms (General disorders) | 0 | 1
Creatinine increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Tremor (Nervous system disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 — Rotator cuff tendinopathy
Abdominal pain (Gastrointestinal disorders) | 1 | 0 — epigastric pain
Non-cardiac chest pain (General disorders) | 1 | 0 — Chest tightness
Abdominal infection (Infections and infestations) | 1 | 0 — diverticular abscess
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 — Aphthous ulcer
Sinusitis (Infections and infestations) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Chest pain (Cardiac disorders) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 — thrush
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1 — elbow pain
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1 — hypersensitivity reaction
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 — superior vena cava occlusion
Lipase increased (Investigations) | 0 | 1
Fever (General disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was stopped prematurely because of slow accrual, leasing to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT02521051/Prot_SAP_000.pdf
  • Informed Consent Form: Phase 1 consent (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02521051/ICF_001.pdf
  • Informed Consent Form: Phase 2 consent (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02521051/ICF_002.pdf